CLINICAL TRIAL: NCT05287425
Title: The Effect of Antibiotic Eye Drops on the Nasal Microbiome in Healthy Subjects, a Phase II Study
Brief Title: The Effect of Antibiotic Eye Drops on the Nasal Microbiome in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Doreen Schmidl, Assoc. Prof. PD, MD, PhD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-240518
Record Dates: First submitted 2021-12-29; First posted 2022-03-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-03

CONDITIONS: Nasal and Pharyngeal Microbiome
MeSH Terms: interventions — Povidone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Gentamicin eye drops (Experimental): 4 drops daily in both eyes for 7 ± 1 days
  Interventions: Drug: Gentamicin Ophthalmic
- Ciprofloxacin eye drops (Experimental): 4 drops daily in both eyes for 7 ± 1 days
  Interventions: Drug: Ciprofloxacin Ophthalmic
- Povidone eye drops unpreserved (Active Comparator): 4 drops daily in both eyes for 7 ± 1 days
  Interventions: Drug: Povidone Ophthalmic
- Povidone eye drops preserved (Active Comparator): 4 drops daily in both eyes for 7 ± 1 days
  Interventions: Drug: Povidone and Benzalkonium Chloride Ophthalmic

INTERVENTIONS:
Drug: Gentamicin Ophthalmic — 4 drops daily in both eyes for 7 ± 1 days
  Arms: Gentamicin eye drops
Drug: Ciprofloxacin Ophthalmic — 4 drops daily in both eyes for 7 ± 1 days
  Arms: Ciprofloxacin eye drops
Drug: Povidone Ophthalmic — 4 drops daily in both eyes for 7 ± 1 days
  Arms: Povidone eye drops unpreserved
Drug: Povidone and Benzalkonium Chloride Ophthalmic — 4 drops daily in both eyes for 7 ± 1 days
  Arms: Povidone eye drops preserved

SUMMARY:
Ophthalmic topical antibiotics are commonly prescribed in clinical practice for several indications such as bacterial conjunctivitis, keratitis, blepharitis, dacryocystitis and also as prophylaxis. Aminoglycosides (i.e. gentamicin) and fluoroquinolones (i.e. ciprofloxacin) are among the most frequently used substance classes.

There is evidence that topical non-antibiotic eye drops might have an effect on the nasopharyngeal mucosal flora. This seems logical due to the anatomical connection through the nasolacrimal duct and the fact that up to 80% of topically administered drug diffuse into the systemic circulation through the highly vascularized nasopharyngeal mucosa. However, in the literature no data on the effect of antibiotic eye drops on the nasal or pharyngeal microbiome are currently available.

Recently, new, non-culture based techniques for assessment of the bacterial microbiome have been developed, so-called "next-generation sequencing" (NGS). NGS utilizes universal primers targeting the 16S rRNA gene, which is ubiquitous across most bacteria. With this technique, it is possible to gain information about a wide range of the bacterial microbiome and not only on pre-selected species.

In the present study, NGS will be used to investigate the effect of antibiotic eye drops on the nasal and pharyngeal microbiome. For this purpose, healthy subjects will be randomized to either receive eye drops containing gentamicin, ciprofloxacin or topical lubricants as control. As secondary outcome, prevalence of bacterial resistance genes, as well as signs and symptoms of ocular surface damage will be assessed.

The study will be carried out in 2 parts. Since both formulations of topical antibiotics contain benzalkonium chloride which also has a potential effect on the nasal and pharyngeal mucosal flora, it is unknown how much benzalkonium chloride would contribute to changes in the nasal microbiome after administration of topical antibiotics. To overcome this problem, first a pilot study in 20 subjects will be performed in which subjects will be randomized to receive either eye drops containing gentamicin, ciprofloxacin, preservative-containing topical lubricants or preservative-free topical lubricants. Based on the results of this pilot study, the control for the main part of the study will be chosen, depending on the effect on the bacterial microbiome. The results of the pilot study could also provide useful data to adjust the sample size for the main study part. In the main study, 60 subjects will be randomized to receive gentamicin, ciprofloxacin or lubricant eye drops. The same examinations as described above will be performed after 1 week treatment as well as 1 week and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 45 years
* Normal ophthalmic findings
* Tear Break Up Time >10 seconds
* Schirmer I Test > 10mm/5min
* Ametropia ≤ 6 diopters
* No use of topical eye or nasal drops in the last 3 months

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages or drugs
* Participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug (except intake of hormonal contraceptives)
* Treatment with topical or systemic antibiotics within 8 weeks before inclusion
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with distribution, metabolism or excretion of study drugs
* Known hypersensitivity to any of the components of the IMP under investigation or other study medication
* Pregnant or breast-feeding women
* Women of childbearing potential (neither menopausal, nor hysterectomized, nor sterilized) not using effective contraception (i.e. oral contraceptives, intra-uterine device, contraceptive implant or condoms)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Nasal bacterial microbiome | change after 1 week treatment
  16S rRNA gene sequencing

SECONDARY OUTCOMES:
Pharyngeal bacterial microbiome | change after 1 week treatment
  16S rRNA gene sequencing
Antibiotic resistance gene prevalence | change after 1 week treatment
Minimum inhibitory concentrations for gentamicin and ciprofloxacin | change after 1 week treatment
Tear film thickness | change after 1 week treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No